CLINICAL TRIAL: NCT03428607
Title: Phase II, Single-arm Study of AZD6738 and Olaparib Combination Therapy in Relapsed Small Cell Lung Cancer Patients [SUKSES-N2]
Brief Title: Study of AZD6738 and Olaparib Combination Therapy in Relapsed Small Cell Lung Cancer Patients [SUKSES-N2]
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Samsung Medical Center (Other)
Responsible Party: Principal Investigator, Keunchil Park, MD, Ph.D, Professor/Director, Samsung Medical Center
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 2017-10-074
Record Dates: First submitted 2018-02-05; First posted 2018-02-09 (Actual); Last update posted 2021-02-18 (Actual); Status verified 2021-02

CONDITIONS: SCLC
MeSH Terms: interventions — ceralasertib; olaparib

STUDY DESIGN:
Oversight: FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: Yes

ARMS (1):
- AZD6738+Olaparib (Experimental): AZD6738 160mg QD per os administered for 7 days and olaparib 300mg BID per os administered daily. One cycle is considered of 28 days.
  Interventions: Drug: AZD6738; Drug: Olaparib

INTERVENTIONS:
Drug: AZD6738 — AZD6738 160mg QD
Drug: Olaparib — Olaparib 300mg BID

SUMMARY:
This study is a single arm, multi-center phase II study of AZD6738 and olaparib combination therapy in patients with relapsed small cell lung cancer (SCLC) as a second or third line chemotherapy.

Patients will receive AZD6738 and olaparib combination therapy. The arm is composed of 45 patients.

AZD6738 160mg QD per os administered for 7 days and olaparib 300mg BID per os administered daily. One cycle is considered of 28 days.

Tumour evaluation using RECIST 1.1 will be conducted at screening (within 28 days prior to first dose) and every 8 weeks relative to the date, up to week 56, then every 12 weeks until objective disease progression (within a window of ± 7 days of the scheduled date).

Study treatment will be continued until objective disease progression (unless other criteria for treatment discontinuation are met). Patients may continue AZD6738 and olaparib beyond progression (according to RECIST 1.1), at the discretion of the investigator if they are clinically benefiting from the treatment and they do not meet any other discontinuation criteria.

If a patient discontinues study treatment prior to disease progression, they should continue to be assessed using RECIST 1.1 until disease progression and then followed up for survival.

Assessments for survival should be made every 8 weeks following objective disease progression. The details of first and subsequent therapies for cancer, after discontinuation of AZD6738 and olaparib treatment, will be collected.

The imaging modalities used for RECIST 1.1 assessment will be CT or MRI scans of chest, abdomen and pelvis. RECIST 1.1 scans will be analysed by the investigator on site.

Patients may also be requested to provide tumour samples from the primary or metastatic tumours on progression to understand resistance mechanisms. Sample provision is optional and depend on the patient's will.

ELIGIBILITY:
Inclusion Criteria:

1. Provision of fully informed consent prior to any study specific procedures.
2. Subjects must be ≥20 years of age.
3. Small cell lung cancer(SCLC) that has progressed during or after first-line therapy.

   * The 1st line regimen must have contained platinum based regimen.
   * Refractory to first-line chemotherapy or relapse within 6 months since the last dose of first-line chemotherapy
   * If the patient correspond to sensitive relapse (relapse more than 6 months since the last dose of first-line chemotherapy), she/he should get second-line treatment.
4. Provision of tumor sample (from either archival or fresh biopsy)
5. Subjects are willing and able to comply with the protocol for the duration of the study including undergoing treatment and scheduled visits and examinations including follow up.
6. ECOG performance status of 0-2
7. Subjects must have a life expectancy ≥ 3 months from proposed first dose date.
8. Subjects must have acceptable bone marrow, liver and renal function measured within 28days prior to administration of study treatment as defined below:

   * Haemoglobin ≥10.0 g/dL with no blood transfusion the past 28days.
   * Absolute neutrophil count (ANC) ≥ 1.5 x 109/L
   * White blood cells (WBC) ≥ 3 x 109/L
   * Platelet count ≥100 x 109/L
   * Total bilirubin ≤ 1.5 x institutional upper limit of normal (ULN) except for subject with liver metastases for whom total bilirubin is ≤ 3 x ULN
   * AST(SGOT)/ALT(SGPT) ≤ 2.5 x institutional upper limit of normal(ULN) except for subject with liver metastases for whom AST(SGOT)/ALT(SGPT) is ≤ 5x ULN
   * Alkaline phosphatase(ALP) ≤ 2.5 x institutional upper limit of normal(ULN) except for subject with liver metastases for whom ALP is ≤ 5 x ULN. ALP is not exclusionary if due to the presence of bone metastasis and liver function is otherwise considered adequate in the investigator's judgement.
   * Subjects must have creatinine clearance estimated using the Cockcroft-Gault equation of ≥51 mL/min:

   Estimated creatinine clearance = (140-age [years]) x weight (kg) x Fa serum creatinine (mg/dL) x 72 a where F=0.85 for females and F=1 for males.

   - Albumin ≥ 33g/L
9. At least one measurable lesion that can be accurately assessed by imaging or physical examination.
10. Evidence of non-childbearing status for women of childbearing potential: A woman of childbearing potential must have a negative or urine pregnancy test at screening and confirmed prior to treatment on Cycle 1 Day 1
11. Female subjects who are not of childbearing potential and fertile female subjects of childbearing potential who agree to use adequate contraceptive measures, who are not breastfeeding. For women, must agree to use a barrier method of birth control. must agree to use a barrier method of birth control for 3months after treatment stops.
12. Fertile male patients willing to use at least one medically acceptable form of birth control, and must not donate sperm, for the duration of the study, and for 6months after treatment stops.
13. Provision of informed consent for genetic research. If a patient declines to participate in the genetic research, there will be no penalty or loss of benefit to the patient. The patient will not be excluded from other aspects of the study described in this Clinical Study Protocol, so long as they consent to that part.

Exclusion Criteria:

1. Previous enrolment in the present study
2. More than two prior chemotherapy regimen for the treatment of small cell lung cancer
3. Any previous treatment with ATR inhibitor and PARP inhibitor, including olaparib
4. Patients with second primary cancer, except: adequately treated non-melanoma skin cancer, curatively treated in-situ cancer of the cervix, or other solid tumours curatively treated with no evidence of disease for >2 years.
5. Subjects unable to swallow orally administered medication.
6. Treatment with any investigational product during the last 14 days before the enrollment (or a longer period depending on the defined characteristics of the agents used).
7. Subjects receiving any systemic chemotherapy, radiotherapy (except for palliative reasons), within 2 weeks from the last dose prior to study treatment The patient can receive a stable dose of bisphosphonates or denosumab for bone metastases, before and during the study as long as these were started at least 4 weeks prior to treatment.
8. Concomitant use of known sensitive CYP3A4 substrates or CYP3A4 substrates with a narrow therapeutic index, or to be moderate to strong CYP3A4 inhibitor/inducer which cannot be discontinued to 2weeks prior to Day 1 of dosing(except for St. John's Wort, which is 3 weeks) and withheld throughout the study until 4weeks after the last dose of study drug, Co-administration of aprepitant or fosaprepitant or Pgp inhibitor/inducer during this study is prohibited Refer to the Section 8.3.2 and Appendix H for listing of all prohibited medications.
9. With the exception of alopecia, any ongoing toxicities (>CTCAE 4.03 grade 1) caused by previous cancer therapy.
10. Intestinal obstruction or CTCAE 4.03 grade 3 or grade 4 upper GI bleeding within 4weeks before the enrollment.
11. Subjects with myelodysplastic syndrome/acute myeloid leukemia or with features suggestive of MDS/AML.
12. Resting ECG with measurable QTc > 470 msec on 3 or more time points within a 24 hour period or any factors that increase the risk of QTc prolongation or risk of arrhythmic events such as heart failure, hypokalaemia, congenital long QT syndrome, immediate family history of long QT syndrome or unexplained sudden death under 40 years of age.
13. Subjects with cardiac problem as follows: unstable angina pectoris, congestive heart failure, acute myocardial infarction, conduction abnormality not controlled with pacemaker or medication, significant ventricular or supraventricular arrhythmias (patients with chronic rate controlled atrial fibrillation in the absence of other cardiac abnormalities are eligible).
14. Subjects at risk of brain perfusion problems(e.g., carotid stenosis hypotension, including a fall in blood pressure of >20mm Hg)
15. Subjects with relative hypotension (< 100/60 mm Hg) or clinically relevant orthostatic
16. Uncontrolled hypertension requiring clinical intervention.
17. Female patients who are breast-feeding or child-bearing
18. Any evidence of severe or uncontrolled systemic disease, active infection, active bleeding diatheses or renal transplant, including any subjects known to have human immunodeficiency virus (HIV), active hepatitis B or active hepatitis C
19. Major surgical procedures ≤28 days of beginning study treatment, or minor surgical procedures ≤7 days
20. Known central nervous system (CNS) disease other than neurologically stable,treated brain metastases - defined as metastasis having no evidence of progression or haemorrhage for at least 2weeks after treatment.

Min Age: 20 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 26 (Actual)
Dates: Start 2018-10-17 (Actual); Primary Completion 2021-01-15 (Actual); Study Completion 2021-01-15 (Actual)

PRIMARY OUTCOMES:
Objective response rate (ORR) by RECIST 1.1 | up to 18 months
  Assessments to be performed using CT or MRI scans. to be measured

SECONDARY OUTCOMES:
Duration of response | up to 18 months
  Assessments to be performed using CT or MRI scans. to be measured
Disease control rate | At 8 weeks
  Assessments to be performed using CT or MRI scans. to be measured
Overall survival | up to 18 months
  Kaplan-Meier method
progression-free survival | up to 18 months
  Kaplan-Meier method
Time to first relapse | up to 18 months
  Assessments to be performed using CT or MRI scans. to be measured

CONTACTS AND LOCATIONS:
Locations (1):
- Samsung Medical Center, Seoul, South Korea